## Statistical analysis plan

Title: Effect of Structured Progressive Task-Oriented Circuit Class Training

With Motor Imagery on Gait in Stroke

Clinical registration

no:

NCT03436810

**Documentt date:** January 18, 2017

## Statistical analysis plan:

All data will be tested by the SPSS version 18.0 with a significant value of p < 0.05 for all comparisons. The demographic data of the participants will be presented with mean, standard deviation, and range for the continuous variables. Frequency and percentage will be presented for the categorical variables.

Normality will be tested by the Kolmogorov Smirnov Goodness of Fit test, for normally distributed variables, a two-way mixed repeated measure ANOVA will be tested to investigate the effect of group and time on the outcome measures. In addition, the interaction effect of the group by time will be detected. For the non-normally distributed variables, the Mann-Whitney U test (betweengroup) and the Friedman ANOVA test in conjunction with the Wilcoxon Signed-Rank test (withingroup) will be used.